CLINICAL TRIAL: NCT02175355
Title: A Randomised, Double- Blind, Placebo-controlled, 6 Week Parallel-group Trial on the Efficacy and Safety of the Angiotensin II Receptor Antagonist Micardis® (Telmisartan 20 mg, 40 mg or 80 mg, p.o. Once Daily) or Hydrochlorothiazide 12.5 mg p.o. Once Daily in the Management of Patients With Isolated Systolic Hypertension (ISH). (ARAMIS - Study = Angiotensin II Receptor Antagonist Micardis in Isolated Systolic Hypertension)
Brief Title: Efficacy and Safety of the Angiotensin II Receptor Antagonist Micardis® (Telmisartan) or Hydrochlorothiazide in the Management of Patients With Isolated Systolic Hypertension (ISH)
Acronym: ARAMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.254
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

ARMS (5):
- Low dose of Micardis® (Experimental)
  Interventions: Drug: Low dose of Micardis®
- Medium dose of Micardis® (Experimental)
  Interventions: Drug: Medium dose of Micardis®
- High dose of Micardis® (Experimental)
  Interventions: Drug: High dose of Micardis®
- Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of Micardis®
  Arms: Low dose of Micardis®
Drug: Medium dose of Micardis®
  Arms: Medium dose of Micardis®
Drug: High dose of Micardis®
  Arms: High dose of Micardis®
Drug: Hydrochlorothiazide
  Arms: Hydrochlorothiazide
Drug: Placebo
  Arms: Placebo

SUMMARY:
Primary: To identify doses of Micardis®(telmisartan) which, administered once daily, are more effective than placebo and not inferior to HCTZ in lowering systolic blood pressure (SBP) in patients with isolated systolic hypertension (ISH), and to assess the dose response relationship of the antihypertensive effect of telmisartan over the dose range of 20 to 80 mg.

Secondary: Target fall in SBP, change from baseline in seated DBP. Safety and tolerability of Micardis® and HCTZ in patients with ISH as measured by changes in physical examinations, heart rate, laboratory parameters and/or 12-lead ECG, as well as the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years, but less than 85 years of age
* Mean SBP ≥ 150 mm Hg and mean DBP < 90 mm Hg at the randomisation visit (visit 2), according to WHO definitions of ISH (excluding the subgroup of borderline ISH)
* Hypertensive patients not on current antihypertensive therapy or able to stop current treatment for a period of up to 8 - 10 weeks without endangering the health of the patient (investigator's discretion)
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to start of run-in period) who:

  1. are not surgically sterile; and/or
  2. are nursing
  3. are of child-bearing potential and are not practicing acceptable means of birth control or do NOT plan to continue using this method throughout the study. Acceptable methods of birth control include oral, implantable or injectable contraceptives
* Mean systolic blood pressure ≥ 180 mmHg at the randomization Visit 2
* Known or suspected secondary hypertension
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  1. Serum glutamic pyruvate transaminase (ALT) or serum glutamic oxaloacetic transaminase (AST) > than 2 times the upper limit of normal range
  2. Serum creatinine > or 1.8 mg/dl (or 159 µmol/l)
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney, patients post-renal transplant or with only one functioning kidney
* Clinically relevant hypokalemia or hyperkalemia
* Uncorrected volume or sodium depletion
* Primary aldosteronism
* Hereditary fructose intolerance
* Biliary obstructive disorders
* Symptomatic congestive heart failure
* Angina pectoris or previous myocardial infarction
* Previous percutaneous transluminal coronary angioplasty or coronary artery bypass craft
* Previous cerebrovascular accident or hypertensive encephalopathy or transient ischemic attack(s)
* Current treatment with any antihypertensive agents, whether or not prescribed for this indication, that cannot be safely stopped (investigators decision) by the start of the run-in period. Any pre-treatment with diuretics, ACE inhibitors or angiotensin II receptor antagonists requires an extension of the run-in period from 2 to 4 weeks for adequate wash-out
* Atrial fibrillation (controlled or otherwise) or any other clinically relevant cardiac arrhythmias as determined by the clinical investigator
* Hemodynamically relevant aortic or mitral valve stenosis, obstructive hypertrophic cardiomyopathy or other outflow obstruction of the left ventricle
* Patients with non-insulin-dependent diabetes mellitus requiring treatment with oral hypoglycemics who fail to meet the following criteria by history:

  1. Fasting blood glucose less than 200 mg/dl (11.1 mmol/l)
  2. Therapy stabilized for at least one month prior to start of placebo run-period
* Patients with diabetes mellitus requiring treatment with insulin
* Patients who have previously experienced symptoms characteristics of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists
* Known drug or alcohol dependency
* Any investigational therapy within one month of signing the informed consent form and during the trial
* Known hypersensitivity to any component of the formulation of telmisartan or hydrochlorothiazide including allergy to sulfonamides
* Concomitant use of lithium or cholestyramine or colestipol resins (potential drug interactions with HCTZ)
* Gout (contraindication for treatment with HCTZ)
* Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of telmisartan or hydrochlorothiazide

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 1999-10; Primary Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated systolic blood pressure at trough (24 hours post-dose) | after 6 weeks of treatment
Change from baseline in urine albumine excretion rate | after 6 weeks of treatment
Change from baseline in pulse wave velocity | after 6 weeks of treatment

SECONDARY OUTCOMES:
Percentage of patients achieving a target fall in SBP | after 6 weeks of treatment
Changes in seated diastolic blood pressure (DBP) | up to 6 weeks
Change from baseline in augmentation index | after 6 weeks of treatment
Incidence and intensity of adverse events | up to 6 weeks
Number of patients with relevant changes from baseline in physical examination | baseline, week 6
Number of patients with relevant changes in Heart Rate (HR) | up to 6 weeks
Number of patients with relevant changes in laboratory parameters | up to 6 weeks
Number of patients with relevant changes in 12-lead electrocardiogram (ECG) | up to 6 weeks